CLINICAL TRIAL: NCT00492141
Title: Aerosol Liposomal 9-Nitro-20(S)-Camptothecin (L9-NC) and Temozolomide in Ewing's Sarcoma and Other Solid Tumors With Lung Involvement
Brief Title: Aerosol L9-NC and Temozolomide in Ewing's Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0889
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Ewing's Sarcoma
Keywords: Ewing's Sarcoma; Lung Involvement; Temozolomide; Temodar; Aerosol Liposomal 9-Nitro-20(S)-Camptothecin; Aerosol L9-NC; L9-NC
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Temozolomide; rubitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L9-NC + Temozolomide (Experimental): Liposomal 9-nitro-20(S)-camptothecin (L9-NC) alone, total 10 ml of 0.4 mg/ml in aerosol reservoir once a day for 5 days in row each 2 weeks, followed by 2 weeks off; then in combination with Temozolomide 100 mg/m^2 oral/day for Cycle 2 Days 1-5.
  Interventions: Drug: Temozolomide; Drug: L9-NC

INTERVENTIONS:
Drug: Temozolomide — Cycle 2, Dose Level 1 = 100 mg/m^2 by mouth (PO) Daily, Days 1-5 Prior to L9-NC; Cycle 3, Dose Level 2 = If the patient has no toxicity greater than grade 2, advance to 100 mg/m^2 PO Every 12 Hours, Days 1-5 Prior to L9-NC. If the patient is not able to advance to dose level 2, the patient may continue at dose level 1 as in cycle 2; Cycle 4 and beyond = Patients will continue on dose level 1 or 2 as given in cycle 3.
  Other Names: Temodar
Drug: L9-NC — Cycle 1 = Administered by aerosol 5 consecutive days per week for 2 weeks. A total of 10 ml of 0.4 mg/ml in an aerosol reservoir delivered over approximately 30 minutes per day given once a day, 5 days a week, for 2 weeks, followed by 2 weeks off.
  Cycle 2, Dose Level 1 = Week 1, doses 1-5 preceded by temozolomide. Continue L9-NC once a day, 5 days a week, for 2 weeks, followed by 2 weeks off.
  Cycle 3, Dose Level 2 = If the patient has no toxicity greater than grade 2, due to drug, during cycle 2, L9-NC may be increased to twice daily, approximately 12 hours apart. Week 1, the morning dose on days 1-5 preceded by temozolomide. L9-NC will be given twice a day, 5 days a week, for 2 weeks, followed by 2 weeks off. If the patient is not able to advance to dose level 2, the patient may continue at dose level 1 as in cycle 2.
  Cycle 4 and beyond, patients will continue on dose level 1 or 2 as given in cycle 3.
  Other Names: 9-Nitro-20(S)-Camptothecin; Aerosol L9-NC

SUMMARY:
Primary Objectives:

1. To determine the feasibility and toxicity profile of administering liposomal 9-Nitro-20-(S)-Camptothecin (L9-NC) by aerosol alone and in combination with temozolomide.
2. To determine the effectiveness of L9-NC given by aerosol in combination with temozolomide in patients with solid tumors involving the lungs.

DETAILED DESCRIPTION:
L9-NC and temozolomide each work by blocking certain tumor cell functions, which can keep tumor cells from growing.

If you are found to be eligible to take part in this study, you will be given the L9-NC aerosol (an inhaled spray) by mouth through a face mask for Cycle 1 of therapy. You will receive L9-NC over about 30 minutes once a day, for 5 days in a row. This will be done for 2 weeks. Doctors will then monitor you for safety for another 2 weeks after treatment. A treatment cycle lasts for 4 weeks.

Your first L9-NC aerosol treatment, during Cycle 1, will be given at M.D. Anderson. You may receive the rest of your treatments at home, if you experienced no bad side effects with the first aerosol treatment.

During Cycle 2 of therapy, if you have not experienced any intolerable side effects, you will be given temozolomide. You will receive temozolomide by mouth once a day, for 5 days in a row, during the first week of each cycle. You will also continue to receive the L9-NC aerosol over about 30 minutes once a day, for 5 days in a row, for 2 weeks. Doctors will then monitor you for safety for another 2 weeks after treatment.

During Cycle 3 of therapy, if you have not experienced any intolerable side effects, you will continue to be given temozolomide by mouth once a day, for 5 days in a row, during the first week of each cycle. You will receive the L9-NC aerosol twice a day, about 12 hours apart, over about 30 minutes, for 5 days in a row, for 2 weeks. If you experience any bad side effects during Cycle 2, your dose of temozolomide will be decreased, and you will continue to receive L9-NC aerosol once a day (instead of twice a day), for 5 days in a row, for 2 weeks.

For all further cycles of treatment, if you experienced any bad side effects during Cycle 3, you will receive L9-NC only once a day, instead of twice a day. If you are already receiving L9-NC only once a day, and you experience intolerable side effects in Cycle 3, you will be taken off this study.

You will be shown how to do spirometry (a lung test that measures how much and how fast air moves out of the lungs) to monitor the safety of your therapy. You will be asked to do this after each treatment cycle, for the first 2 cycles. If your dose of L9-NC is increased to twice a day, you will also be asked to do spirometry after the second dose of the day during Cycle 3. For future cycles, you will be asked to do spirometry after the last dose of L9-NC, on the first day of each week of treatment. The results of spirometry will need to be sent to M.D. Anderson by telephone, after each test. The results will be sent electronically. They will be reviewed every day after they are received, and you will be contacted if there are abnormal results. Your doctor may also perform additional spirometry as needed.

You will be examined by a doctor before the second and third cycle of therapy (every 4 weeks). You will have blood drawn (about 2 tablespoons) every week during the first 2 to 3 cycles of therapy. After Cycle 3 of therapy, blood tests (about 2 tablespoons) will be done before each cycle of therapy. Chest x-rays, CT chest scans, and any other imaging studies, as done at the beginning of this study, will be done to measure your disease and will be repeated after every 3 cycles of therapy. You will also have a breathing function test, if the doctor thinks it is necessary.

If your tumor size decreases during this treatment, you may have other therapy performed, such as surgery, radiation, or radiofrequency ablation, outside of this study. If the treatment in this study alone, or in combination with other therapy, results in complete disappearance of your disease, your treatment on this study may continue for up to 6 more cycles.

You will be taken off this study if your disease gets worse or you experience any intolerable side effects. If you are taken off this study for intolerable side effects, you will be followed-up for 30 days after treatment ends or until your side effects go away.

If you have a complete remission, chest x-rays, CT chest scans, and any other imaging studies, as done at the beginning of this study, will be done to look for disease about every 3 months after completion of treatment.

This is an investigational study. L9-NC is authorized by the FDA for use in research only. Temozolomide is approved by the FDA. The use of these drugs together in this study is experimental. Up to 40 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 10 years of age or older, with primary or metastatic cancer in the lungs, who have failed or progressed on front line therapy and have no standard therapies available for treatment are eligible. Patients may also have disease in other sites, but must have current lung involvement to be eligible.
* Patients should have adequate bone marrow function, defined by: absolute peripheral granulocyte count of >/= 1500 cells/mm^3, platelet count > 100,000 platelets/mm^3, and Hgb > 8.0 g/dl. For patients with documented bone marrow involvement, the following counts are acceptable for enrollment: absolute peripheral granulocyte count of > 1000 cells/mm^3 , platelet count > 75,000 platelets/mm^3.
* Patients should have adequate hepatic function, defined by: total bilirubin < 2 mg/dl and ALT or AST < 2x upper limit of normal.
* Patients should have adequate renal function, defined by serum creatinine </= 2 mg/dl.
* Patients must have adequate pulmonary function, as defined by a pulmonary function test with: >/= 50% FVC, >/= 50% FEV1 and >/= 50% DLCO of predicted values

Exclusion Criteria:

* Patients with symptomatic brain metastases.
* Pregnant women or nursing mothers. Patients of child bearing potential must use adequate contraception.
* Patients receiving concurrent chemotherapy.
* Patients may not receive concurrent radiation therapy to the chest during cycles 1-3. Radiation therapy to disease in other areas of the body is permissible at any time, but such lesions will not be evaluable for response. Although patients who have received prior radiation to the chest are eligible, patients should be at least 4 weeks from prior radiation to the chest. Any chest lesion treated with radiation must have progressed to be considered measurable for this study.
* Patients with severe medical problems such as uncontrolled diabetes mellitus (glucose consistently greater than 200 mg/dl, or Hemoglobin A1c greater than 8%) or symptomatic cardiovascular disease (New York class III) or active infections requiring IV antibiotics are not eligible for this trial.
* Patients requiring oxygen.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Toxicity Profile | From baseline to end study period (3 years)
  Toxicity profile of administering liposomal 9-Nitro-20-(S)-Camptothecin (L9-NC) by aerosol alone and in combination with temozolomide. All toxicities evaluated according to NCI Common Toxicity Criteria, Version 3.0 and recorded prior to each cycle of therapy.

SECONDARY OUTCOMES:
Number of Participants with Response According to Response Evaluation Criteria In Solid Tumors (RECIST) | Baseline till after three cycles of therapy (approximately 9 weeks)
  Response by tumor measurements (centimeters) using RECIST criteria: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): >20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of one or > new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E. Herzog, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org